CLINICAL TRIAL: NCT02114515
Title: PATient Navigator to rEduce Readmissions
Acronym: PArTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Society of Hospital Medicine (Other); COPD Foundation (Other); University of Kentucky (Other); Mended Hearts (Unknown); American Heart Association (Other); Sickle Cell Disease Association of Illinois (Unknown); AcademyHealth (Other); The National Association of Social Workers Foundation (Unknown); Respiratory Health Association (Unknown); University of Illinois Sickle Cell Patient Council (Unknown); National Jewish Health (Other); Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Jerry Krishnan, Professor of Medicine and Public Health; Associate Vice Chancellor for Population Health Sciences, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PCORI-IH 1211-4365
Record Dates: First submitted 2014-04-01; First posted 2014-04-15 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Heart Failure; Sickle Cell Disease; Myocardial Infarction; Pneumonia
Keywords: Patient Navigators; Readmissions; Peer Coaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Anemia, Sickle Cell; Myocardial Infarction; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Hospital usual care
  Hospital usual care: Written discharge instructions provided to patients prior to hospital discharge.
  Interventions: Behavioral: Hospital usual care
- Usual Care + PArTNER (Experimental): Navigator intervention: (Community health worker, peer-led telephone support line, usual care)
  Hospital usual care: Written discharge instructions provided to patients prior to hospital discharge.
  Community health worker: The community health worker provides social support, literacy appropriate education, and acts as a conduit between the patient and the patient's medical team
  Peer-led telephone support line: The peer-led telephone support line will provide social support, peer-to-peer coaching, and facilitate communication with the patient's medical care team.
  Interventions: Behavioral: Hospital usual care; Behavioral: Navigator intervention; Behavioral: Peer-led telephone support line

INTERVENTIONS:
Behavioral: Hospital usual care — Written discharge instructions provided to patients prior to hospital discharge.
Behavioral: Navigator intervention — A Patient Navigator will provide social support, literacy appropriate education, and act as a conduit between the patient and the patient's medical team
  Arms: Usual Care + PArTNER
Behavioral: Peer-led telephone support line — The peer-led telephone support line will provide social support, peer-to-peer coaching, and facilitate communication with the patient's medical care team.
  Arms: Usual Care + PArTNER

SUMMARY:
Staying out of the hospital is valued by patients and their caregivers. Their interests converge with those of hospitals now that high 30-day readmission rates for some conditions place hospitals at risk for financial penalties from the Centers for Medicare and Medicaid Services. This study focuses on developing and testing a program that combines a community health worker (lay patient advocate, acting as a "Patient Navigator") and a peer-led telephone support line to improve patient experience during hospital to home transition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older on date of hospital admission
2. Hospitalized at the University of Illinois Hospital, Chicago
3. Admission diagnosis, per treating physician, of pneumonia, COPD, sickle cell disease, heart failure, or myocardial infarction
4. Receive medical care on an inpatient medical service

Exclusion Criteria:

1. Unable to understand and speak English
2. Unable/decline to give informed consent
3. Previous participant in PArTNER
4. Planned transfer to another acute care facility
5. Planned discharge to facility other than home (e.g. long term care facility)
6. Currently on hospice or plans to discharge home to hospice
7. Current plans to leave against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Krishnan, MD, PhD, Principal Investigator — University of Illinois at Chicago; Elizabeth Calhoun, PhD, Principal Investigator — University of Arizona; Mark V. Williams, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Illinois Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] LaBedz SL, Prieto-Centurion V, Mutso A, Basu S, Bracken NE, Calhoun EA, DiDomenico RJ, Joo M, Pickard AS, Pittendrigh B, Williams MV, Illendula S, Krishnan JA. Pragmatic Clinical Trial to Improve Patient Experience Among Adults During Transitions from Hospital to Home: the PArTNER study. J Gen Intern Med. 2022 Dec;37(16):4103-4111. doi: 10.1007/s11606-022-07461-0. Epub 2022 Mar 8. PMID 35260961
- See also: Patient-Centered Outcomes Research Institute (PCORI): Funding Award details — http://www.pcori.org/research-results/2013/patient-navigator-reduce-readmissions-partner

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Usual Care + PArTNER
Started | 511 | 518
Completed | 378 | 368
Not Completed | 133 | 150
Not completed — Lost to Follow-up | 52 | 55
Not completed — Death | 12 | 12
Not completed — Withdrawal by Subject | 4 | 22
Not completed — Other | 65 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Usual Care + PArTNER | Total
Number analyzed (Participants) | 511 | 518 | 1029
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 412 | 423 | 835
  >=65 years | 99 | 95 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (17.0) | 49.8 (16.5) | 49.9 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 277 | 567
  Male | 221 | 241 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 49 | 89
  Not Hispanic or Latino | 471 | 468 | 939
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 424 | 423 | 847
  White | 62 | 72 | 134
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 511 | 518 | 1029

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Emotional Distress-Anxiety (v1.0, SF4a)
Description: Change in T-score from baseline to 30 days post discharge (30 days minus baseline).
  A change in t-score <0 indicates improvement. A change equal to 0 indicates no change. A change >0 indicates worsening.
Time Frame: 30 days post discharge
Population: Due to missing data, the number of participants analyzed may be less than the numbers provided in the Participant Flow module.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 406 | 391
T-score | -0.2 (0.5) | -1.7 (0.5)

2. Primary Outcome: PROMIS Informational Support (v2.0, SF4a)
Description: Change in T-score from baseline to 30 days post discharge (30 days minus baseline).
  A change in t-score <0 indicates worsening. A change equal to 0 indicates no change. A change >0 indicates improvement.
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 405 | 391
T-score | 2.3 (0.6) | 2.5 (0.6)

3. Secondary Outcome: PROMIS Emotional Support (v2.0, SF4a)
Description: as for outcome 2
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 401 | 390
T-score | -0.1 (0.5) | -0.1 (0.5)

4. Secondary Outcome: PROMIS Instrumental Support (v2.0, SF4a)
Description: as for outcome 2
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 403 | 391
T-score | 1.0 (0.5) | 0.6 (0.5)

5. Secondary Outcome: PROMIS Global Health, Physical (v1.1, SF)
Description: as for outcome 2
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 408 | 389
T-score | 4.6 (0.4) | 4.4 (0.4)

6. Secondary Outcome: PROMIS Global Health, Mental (v1.1, SF)
Description: as for outcome 2
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 408 | 389
T-score | 0.8 (0.4) | 0.6 (0.4)

7. Secondary Outcome: PROMIS Emotional Distress-Anxiety (v1.0, SF4a)
Description: Change in T-score from baseline to 60 days post discharge (60 days minus baseline).
  A change in t-score <0 indicates improvement. A change equal to 0 indicates no change. A change >0 indicates worsening.
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 375 | 365
T-score | 0.3 (0.6) | -1.1 (0.6)

8. Secondary Outcome: PROMIS Informational Support (v2.0, SF4a)
Description: Change in T-score from baseline to 60 days post discharge (60 days minus baseline).
  A change in t-score <0 indicates worsening. A change equal to 0 indicates no change. A change >0 indicates improvement.
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 373 | 363
T-score | 1.7 (0.6) | 2.0 (0.7)

9. Secondary Outcome: PROMIS Emotional Support (v2.0, SF4a)
Description: as for outcome 8
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 372 | 363
T-score | 0.1 (0.5) | -0.2 (0.5)

10. Secondary Outcome: PROMIS Instrumental Support (v2.0, SF4a)
Description: as for outcome 8
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 374 | 363
T-score | 0.8 (0.5) | 1.0 (0.5)

11. Secondary Outcome: PROMIS Global Health, Physical (v1.1, SF)
Description: as for outcome 8
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 372 | 365
T-score | 3.4 (0.5) | 3.6 (0.4)

12. Secondary Outcome: PROMIS Global Health, Mental (v1.1, SF)
Description: as for outcome 8
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 372 | 366
T-score | -1.3 (0.5) | 01.1 (0.4)

13. Secondary Outcome: Death
Description: Caregiver-reported and confirmed by EHR review
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 502 | 497
Participants | 4 | 7

14. Secondary Outcome: Death
Description: Caregiver-reported and confirmed by EHR review
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 493 | 488
Participants | 9 | 9

15. Secondary Outcome: Re-hospitalization or Death
Description: Confirmed by EHR review
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 503 | 495
Participants | 100 | 112

16. Secondary Outcome: Re-hospitalization or Death
Description: Confirmed by EHR review
Time Frame: 60 days post discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 493 | 487
Participants | 147 | 159

17. Secondary Outcome: ED Visit, Re-hospitalization, or Death
Description: Confirmed by EHR review
Time Frame: 30 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 503 | 495
Participants | 156 | 154

18. Secondary Outcome: ED Visit, Re-hospitalization, or Death
Description: Confirmed by EHR review
Time Frame: 60 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 494 | 487
Participants | 210 | 216

19. Secondary Outcome: Outpatient Healthcare Visit
Description: Self-reported
Time Frame: 14 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 405 | 388
Participants | 137 | 112

20. Secondary Outcome: Outpatient Healthcare Visit
Description: EHR-reported
Time Frame: 14 days post discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care + PArTNER
Number analyzed (Participants) | 511 | 507
Participants | 236 | 232

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through 60 days after hospital discharge.
Arm/Group | Usual Care | Usual Care + PArTNER
All-Cause Mortality (participants affected / at risk) | 12/511 | 12/518
Serious Adverse Events (participants affected / at risk) | 12/511 | 12/518
Other Adverse Events (participants affected / at risk) | 0/511 | 0/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=511) | Usual Care + PArTNER (N=518)
All-cause death (General disorders) | 12 | 12 — Causes of death were not collected.

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No